CLINICAL TRIAL: NCT02086188
Title: Pilot Study of Mirabegron and Behavioral Modification Including Pelvic Floor Exercise for Overactive Bladder in Multiple Sclerosis (MIRROR)
Brief Title: Study of Behavioral Modification Program and Mirabegron to Improve Urinary Urgency in Multiple Sclerosis
Acronym: MIRROR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Theodore R. Brown, MD MPH (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor-Investigator, Theodore R. Brown, MD MPH, Medical Director - MS Neuro-Rehabilitation, EvergreenHealth
Organization: EvergreenHealth (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRB2013
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Results first posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Overactive Bladder; Incontinence; Voiding; Bladder Urgency; Pelvic Floor Exercises
MeSH Terms: conditions — Multiple Sclerosis; Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirabegron (Experimental): Mirabegron - 25mg (one tablet) taken by mouth daily with option to up-titrate to 50mg daily (two tablets) taken by mouth daily
  Interventions: Drug: Mirabegron
- Placebo (Placebo Comparator): Placebo - one tablet taken by mouth daily and two tablets taken by mouth daily if subject chooses up-titration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirabegron — see detailed information in associated Arm Description
  Other Names: MBG; Myrbetriq
  Arms: Mirabegron
Drug: Placebo — Sugar pill manufactured to mimic Mirabegron 25mg tablet.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if treatment with Mirabegron will improve urinary urgency control beyond that achieved with pelvic floor exercises alone

DETAILED DESCRIPTION:
A randomized 1:1 placebo controlled 10-week study of mirabegron as add-on therapy to an educational intervention on behavioral modification including pelvic floor exercise (BM-PFE) to a cohort of 40 Multiple Sclerosis (MS) subjects with overactive bladder (OAB). Trial will last approximately 12 weeks for each subject, including screening period and treatment period.

Active drug will be mirabegron 25mg daily with optional up-titration to 50mg daily after approximately 5 weeks. Subjects will be randomized at the Baseline Visit based on recordings in a voiding diary kept for 72 continuous hours in the screening period.

Voiding diaries of a 72 hour period each will be utilized during the screening period, between Phone Visit 1 and Titration and between Phone Visit 2 and Final Visit. In the diaries, subjects will record the time of each micturition and/or urgency episode, urine volume with each void (when available), any episode of incontinence, and the severity of urgency (Overactive Bladder Symptom Composite Score, mean of 72 hour total daily cumulative score.

Primary outcome will be average daily OAB-SCS total score, Final Visit vs. Baseline. This accounts for the frequency, urgency and incontinence components of OAB.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Multiple Sclerosis (MS) (no sub-type restrictions)
* Age ≥18
* No change in disease modifying therapy in 60 days.
* Patient willing and able to complete micturition diary
* Urinary urgency (8 or more entries of bladder urgency score ≥2) in 72hr voiding diary recorded during screening period
* Micturition frequency ≥ 8 / day or incontinence ≥ 2 episodes in 72 hour voiding diary recorded during screening period
* At least 36 hours of voiding activity recorded in 72 hour voiding diary during screening period
* Non-antimuscarinic medications that are likely to influence bladder function may not be initiated between screening and study completion. They may be continued with no dose changes during the study.
* Discontinued use of antimuscarinics at least two weeks prior to screening
* Able to give informed consent

Exclusion Criteria:

* Females who are breast-feeding, pregnant or have potential to become pregnant during the course of the study (fertile and unwilling/unable to use effective contraceptive measures)
* Multiple Sclerosis exacerbation within 30 days of screening
* Cognitive deficits that would interfere with the subject's ability to give informed consent or perform study testing
* Screening blood pressure > 165 systolic or 100 diastolic
* History of allergy to Mirabegron
* Screening post-void residual > 200ml
* Evidence of urinary tract infection at screening
* Evidence of chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy, or previous or current malignant disease of the pelvic organs
* Intravesical botulinum toxin treatment within the previous six months of screening.
* Presence of InterStim device
* Use of indwelling catheter or self-catheterization
* Concurrent use of thioridazine(Mellaril® or Mellaril-S®, flecainide (Tambocor®), propafenone (Rythmol®) or digoxin (Lanoxin®)
* Concurrent use of antimuscarinics: oxybutynin (Ditropan®, Ditropan XL ®), tolterodine (Detrol®, Detrol LA®), fesoterodine extended-release (Toviaz®), solifenacin (Vesicare®), trospium (Sanctura®, Sanctura XR®), darifenacin extended release (Enablex®)
* Screening estimated glomerular filtration rate (eGFR) < 60, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2x upper limit of normal
* Any other serious and/or unstable medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore R Brown, MD, MPH, Principal Investigator — EvergreenHealth
Locations (1):
- EvergreenHealth MS Center, Kirkland, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mirabegron | Placebo
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirabegron | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Median (Full Range); unit: years] | 55 [35 to 67] | 50 [35 to 82] | 53 [35 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Overactive Bladder Symptom Composite Score (OAB-SCS) at Baseline vs. Final Visit
Description: Primary outcome: Overactive Bladder Symptom Composite Score (OAB-SCS) total score, average daily, Baseline vs. Final Visit The OAB-SCS measures symptoms of overactive bladder, urgency, frequency, incontinence. This is an ordinal scale is 1-5, 1 (minimum) = no urgency, 5 (maximum) = urgency incontinence.
  Higher values represent a worse outcome.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Placebo - one tablet taken by mouth daily and two tablets taken by mouth daily if subject chooses up-titration
  Placebo: Sugar pill manufactured to mimic Mirabegron 25mg tablet. egron group had a worse outcome on this measure.
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 14 | 14
score on a scale | 3.01 (0.48) | 2.56 (0.84)

2. Secondary Outcome: Overactive Bladder Symptom Composite Score (OAB-SCS) at Baseline vs. Titration Visit
Description: Secondary Outcome Measure based on voiding diary: Average daily Overactive Bladder Symptom Composite Score (OAB-SCS) Baseline compared to Titration Visit The OAB-SCS measures symptoms of overactive bladder, urgency, frequency, incontinence. This is an ordinal scale is 1-5, 1 (minimum) = no urgency, 5 (maximum) = urgency incontinence.
  Higher values represent a worse outcome.
Time Frame: 5 weeks
Population: MS patients with overactive bladder
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 14 | 14
score on a scale | 2.8 (0.64) | 2.23 (0.72)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; Test type: Superiority; p = 0.1911, ANCOVA

3. Secondary Outcome: Mean # of Micturitions/Day Based on Voiding Diaries
Description: Secondary Outcome Measure based on voiding diary:
  Baseline vs Final Visit: mean # of micturitions/day
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: micturitions/day
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 14 | 14
micturitions/day | 6.82 (2.2) | 8.72 (3.14)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; Test type: Superiority; p = 0.4271, ANCOVA

4. Secondary Outcome: Mean # of Incontinence Episodes/Day
Description: Secondary Outcome Measure based on voiding diary:
  Baseline vs. Final Visit: Mean # of incontinence episodes/day
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: Incontinence Episodes/Day
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 14 | 14
Incontinence Episodes/Day | 0.7 (1.09) | 1.05 (2.82)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; Test type: Superiority; p = 0.1723, ANCOVA

5. Secondary Outcome: Mean Volume Voided/Micturition
Description: Secondary Outcome Measure based on voiding diary:
  Baseline vs. Final Visit: Mean volume voided/micturition
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: ml/micturition
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 14 | 14
ml/micturition | 356 (153) | 282 (174)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; Test type: Superiority; p = 0.6340, ANCOVA

6. Secondary Outcome: Qualiveen Questionnaire
Description: Secondary Outcome Measures based on the Qualiveen Questionnaire at Final Visit compared to Baseline Qualiveen questionaire is used, including 8 questions about aspects of bladder problems. Each question is rated 0 (not at all)- 4 (extremely). Overall score is averaged (average score per question)
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 14 | 14
score on a scale | 0.96 (0.84) | 0.71 (0.63)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; Test type: Superiority; p = 0.0091, ANCOVA

7. Secondary Outcome: Subject Global Impression (Single Question)
Description: Secondary Outcome Measures based on the Subject Global Impression (single question) at Final Visit compared to Baseline This is a single question: "How would you rate your level of bladder control during the past week?" 1-7 analog scale, 1 = "terrible'" 7 = "delighted."
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 14 | 14
score on a scale | 5.71 (1.14) | 4.86 (1.29)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Mirabegron | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 6/14 | 4/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirabegron (N=14) | Placebo (N=14)
headache (Nervous system disorders) | 1 (1) | 2 (2) — headache
hypertension (Cardiac disorders) | 0 (0) | 1 (1)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
fatigue (Nervous system disorders) | 1 (1) | 0 (0)
urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT02086188/Prot_SAP_000.pdf